CLINICAL TRIAL: NCT03686475
Title: Is Biodentine, as Successful as, Mineral Trioxide Aggregate for Pulpotomy of Primary Molars? A Split Mouth Clinical Trial
Brief Title: Is Biodentine, as Successful as, Mineral Trioxide Aggregate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Youssef Abd Al Gawad, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: regenerative pulpotomoy
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Dental Caries
Keywords: Pulpotomy, Primary molars, Biodentine, MTA.
MeSH Terms: conditions — Dental Caries | interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine pulpotomy (Experimental): Biodentine (Septodont, France) Pulpotomy for primary molars Clinical and radiographic evaluation Follow up at 1,3,6 and 12 months
  Interventions: Other: Biodentine
- MTA pulpotomy (Active Comparator): MTA (Angelus- Londrina, Brazil) Pulpotomy for primary molars . it is fine hydrophilic powder consisting of tricalcium silicate, tricalicum aluminate, tricalcium oxide, silicate oxide and bismuth oxide11.
  It is currently being used in pulpotomy of primary molars with a high rate of success.
  Clinical and radiographic evaluation. Follow up at 1,3,6 and 12 months
  Interventions: Other: MTA pulpotomy

INTERVENTIONS:
Other: Biodentine — pulpotomy for primary molars , clinical and radiographic evaluation at 1,3,6 and 12month
  Other Names: tricalcium silicate cements
  Arms: Biodentine pulpotomy
Other: MTA pulpotomy — MTA pulpotomy
  Arms: MTA pulpotomy

SUMMARY:
: A split-mouth controlled clinical trial was carried out on 21 healthy, three to seven years old children, with 42 pairs (84 molars) of contralateral mandibular primary molars indicated for pulpotomy. One paired tooth in one side was designated to Biodentine (Group 1) and the other side for MTA (Group 2) as a pulp medicament. All pulpotomized teeth were finally restored with stainless steel crowns. Subjects were monitored clinically and radiographically at one, three, six and 12 months.

DETAILED DESCRIPTION:
Study design:

The present study was a split-mouth controlled clinical trial.

Sample size:

A sample size of 21 patients with 42 pairs of molars (84 molars) was determined using online sample size calculator (Sealed envelope.com).

Subjects:

The study population included three to seven years old healthy and cooperative patients who presented at the Pediatric Dental Clinic, Faculty of Dentistry, Cairo University and had two matched bilateral deep carious mandibular primary molars indicated for pulpotomy, that met specific inclusion criteria. Written consent was obtained from the parent/guardian after explaining the full details of the treatment procedure.

The criteria for inclusion in this study were:

* No history of spontaneous pain
* Absence of tenderness to percussion.
* Absence of physiologic or pathologic tooth mobility.
* No clinical evidence of pulpal inflammation or degeneration, such as history of swelling or presence of sinus tract.
* Restorable teeth.
* Absence of radiographic evidence of internal or external root resorption, pulpal calcification, or osseous disease (periapical or furcation infection).

On the other hand, teeth were excluded if:

* Evidence of necrosis after access cavity preparation.
* Hemostasis could not be achieved within three min after direct contact with a wet cotton pellet, prior to material placement.

Matched molars in each pair were randomly designated using computer software (Random.org) to Group 1: which received Biodentine (Septodont, France), or Group 2: which received MTA (Angelus- Londrina, Brazil), as pulp medicament.

Procedures:

Preoperative periapical radiograph using periapical film size two (Speed D Film, Kodak, US) was taken for the molars considered for treatment. Radiographs should be of proper film density and contrast for proper radiographic diagnosis.

The pulpotomy procedure was performed by the same operator. Local anesthesia was induced and rubber dam isolation was performed, followed by caries removal and deroofing of the pulp chamber using a #330 high-speed carbide bur mounted in a water-cooled high speed turbine. The coronal pulp tissue was amputated using a sterile sharp spoon excavator. The pulp chamber was irrigated with normal saline. Pulp hemostasis was achieved using a sterile wet cotton pellet applied for two to three min.

In Group 1: Biodentine was used according to the manufacturer's instructions. A capsule was gently tapped on a hard surface (to diffuse powder); five drops of liquid from the single dose dispenser were poured into the capsule which was placed in a triturator for 30 sec. The mixture was then introduced into the pulp chamber using amalgam carrier until the entire pulp chamber was completely filled.

In Group 2: MTA was used according to the manufacturer's instructions; the powder was mixed with sterile water in a 3:1 powder/water ratio to obtain a thick creamy paste, then placed on the floor of the pulp chamber using a messing gun and compacted against the pulp orifices with a condenser over a moist cotton pellet.

Molars of both groups were finally restored with stainless steel crowns (3M, ESPE, Unitek, US) cemented with GI cement. An immediate postoperative radiograph using periapical film size two was taken.

Clinical and radiographic evaluation:

All treated patients were followed up at one, three, six and 12 months after the pulpotomy for clinical and radiographic evaluation as recommended by the American Academy of Pediatric Dentistry . Independently, two examiners evaluated the teeth clinically and radiographically.

The pulpotomized teeth were judged as clinically successful if they met the following criteria: Absence of sensitivity, pain, tenderness to percussion, abscess, fistula or tooth mobility. Radiographic success was defined if there were normal periodontal ligament space, absence of furcation or periapical radiolucency, absence of internal or external root resorption. Widening of the periodontal ligament was not considered failure in absence of other concurrent pathologies.

ELIGIBILITY:
Inclusion Criteria:

* No history of spontaneous pain

  * Absence of tenderness to percussion.
  * Absence of physiologic or pathologic tooth mobility.
  * No clinical evidence of pulpal inflammation or degeneration, such as history of swelling or presence of sinus tract.
  * Restorable teeth.
  * Absence of radiographic evidence of internal or external root resorption, pulpal calcification, or osseous disease (periapical or furcation infection).

Exclusion Criteria:

* Evidence of necrosis after access cavity preparation.
* Hemostasis could not be achieved within three min after direct contact with a wet cotton pellet, prior to material placement.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
radiographic success | 1 year
  syptom free

CONTACTS AND LOCATIONS:
Overall Officials: Dr Randa Abd El Gawad, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided